CLINICAL TRIAL: NCT07121452
Title: Tele-Sleep OSA: Clinical Effectiveness, Implementation, and Economic Impact of Telehealth Care for Obstructive Sleep Apnea in the Military Health System
Brief Title: Telehealth for Sleep Apnea: Effectiveness, Implementation, and Cost in the Military Health System
Acronym: TS OSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Collaborators: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USUHS.2024-142; HT94252410479 (Other Grant/Funding Number: Congressionally Directed Medical Research Program (CDMRP))
Record Dates: First submitted 2025-07-17; First posted 2025-08-13 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-07

CONDITIONS: Obstructive Sleep Apnea (OSA)
Keywords: sleep; sleep apnea; treatment; telehealth; implementation
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OSA telehealth care (Experimental): Participants randomized to OSA telehealth care will undergo OSA clinical evaluation via secure video conferencing platform; complete diagnostic OSA testing via established home sleep apnea test (HSAT) procedures; receive comprehensive sleep education; and when indicated, initiate PAP therapy via auto-titrating PAP (APAP). The initial consultation and treatment planning visit will take place with a board-certified sleep medicine physician. Ongoing participant education and support will take place via a secure video conferencing platform with a human sleep navigator (likely a certified clinical sleep health educator [CCSH]).
  Interventions: Behavioral: Sleep Navigator
- Private Sector Care (No Intervention): Participants randomized to private sector care will complete outcomes assessments (i.e., self-report questionnaires) with trained study staff and will undergo treatment as usual.

INTERVENTIONS:
Behavioral: Sleep Navigator — Sleep Navigator will provide education, troubleshooting, motivation, and support pertaining to any additional questions or concerns regarding OSA. They will consult closely with the board-certified sleep medicine physician to ensure that participant care needs are met.
  Other Names: MedBridge
  Arms: OSA telehealth care

SUMMARY:
The long-term goal of this research is to improve military health and operational readiness among military service members with sleep disorders. The overall objective of the current study is to 1) determine the clinical effectiveness (non-inferiority) and cost-effectiveness of OSA telehealth care, including a human sleep navigator (vs private sector care), and 2) to perform a formative evaluation of the implementation of the OSA telehealth care intervention within the National Capitol Region (NCR) market. The central hypothesis is that OSA telehealth care including a human sleep navigator is clinically non-inferior to private sector care and also more cost-effective than private sector care. The investigators plan to achieve the objectives via these 3 Specific Aims: Specific Aim 1: To determine the clinical effectiveness (non-inferiority) of OSA telehealth care, relative to private sector care. Hypothesis 1a: Relative to private sector care, OSA telehealth care is non-inferior for achieving PAP adherence (primary endpoint).

Hypothesis 1b: Relative to private sector care, OSA telehealth care is non-inferior for reducing OSA symptoms and for patient satisfaction (secondary endpoints).

Specific Aim 2: To engage participants via qualitative focus groups and conduct a formative evaluation of the implementation of the OSA telehealth care intervention, using a standardized approach based on the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) framework.

Specific Aim 3: To perform a cost-effectiveness analysis of OSA telehealth care from the DHA perspective.

Hypothesis 3: Relative to private sector care, OSA telehealth care is more cost-effective.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a common and costly chronic medical condition that impacts approximately 27% of men and 9% of women in the U.S. and approximately 936 million adults worldwide. Within the military health system (MHS), the prevalence of OSA is approximately 51.2% and rapidly increasing (e.g., from 11 to 333 per 10,000 ADSMs between the years of 2005 and 2019).3 OSA is characterized by repetitive breathing pauses throughout the night, each lasting a minimum of ten seconds, resulting in blood oxygen desaturations and associated cortical arousals during sleep, as the brain tries harder to breathe and obtain needed oxygen. OSA is associated with worsened medical (cardiovascular disease, stroke, metabolic syndromes [including Type 2 diabetes], and premature death) and mental health (depression, anxiety, traumatic stress, substance misuse) outcomes, and worsened quality of life. Beyond these health consequences, OSA is also associated with dramatically increased costs, including both direct treatment costs as well as indirect costs such as increased risk for motor vehicle crash, lost workplace productivity, and costly workplace accidents and errors. The adverse impact of OSA on readiness and deployability for the Armed Services is also extremely costly. Within the context of the MHS, all direct and most indirect costs are borne by the Defense Health Agency (DHA).

The most common treatment for OSA is positive airway pressure (PAP) therapy. PAP involves a small mask that fits over the nose (or mouth and nose) and gently blows air, creating a pneumatic splint that holds the airway open during sleep. When used as prescribed, PAP results in myriad health benefits, including dramatic reductions in sleepiness and risks associated with sleepiness (e.g., motor vehicle crash), as well as improvements in health-related quality of life (HrQOL), memory, blood pressure, other mental and physical health benefits with high military relevance, and reduced costs.

Unfortunately, despite the high prevalence and well-documented consequences of OSA in the MHS, few studies have examined the impact of OSA treatment on clinical and economic outcomes in the MHS.

Within the MHS there is a gross shortage of trained sleep specialist providers and accredited sleep centers. Thus, the demand for sleep medicine specialty care greatly exceeds available supply. As a result, most MHS beneficiaries receive sleep medicine specialty care through the civilian network and TRICARE contracted providers (i.e., standard purchased care). A typical course of OSA private sector care includes multiple billed face-to-face encounters with a sleep medicine physician, in-lab sleep studies, and provision of PAP equipment billed through various third-party durable medical equipment (DME) providers that are also contracted with TRICARE. Given very high volumes, the costs of standard purchased care borne by the DHA are substantial, and quality is variable. Further, patients often struggle to navigate this complex care process that involves multiple providers with suboptimal care coordination (e.g., primary care, specialty care, DME). Optimizing the approach to OSA care is a vital consideration.

In non-MHS samples, OSA telehealth care has demonstrated clinical non-inferiority and enhanced cost-effectiveness relative to OSA in-person care, while also increasing access to care. For example, home sleep apnea testing (HSAT) and auto-titrating positive airway pressure (APAP) have been extensively validated as viable alternatives to attended in-lab diagnostic sleep studies (i.e., polysomnogram [PSG]) and attended in lab therapeutic sleep studies (i.e., manual PAP titration), respectively. In addition, several studies have highlighted the potential role of non-sleep specialists - including non-physician providers - to increase access to OSA care and deliver high quality OSA care. These findings are especially notable given both the major "virtual first" DHA initiative as well as the DHA Quadruple Aim: improved health readiness, better health, better care, and lower cost. Even so, there remain important gaps in knowledge, particularly from the DHA perspective.

Results from this study are expected to be highly generalizable to ADFM and DEERS beneficiaries diagnosed with obstructive sleep apnea (OSA). Given the prevalence of OSA, the investigators aim to be as inclusive as possible to capture a diverse representation of sex, race/ethnicity, and age.

Within the military health system (MHS), the prevalence of OSA is very high and rapidly increasing. OSA is associated with numerous adverse health consequences, dramatically increased economic costs (including both direct treatment costs as well as indirect costs) and reduced military readiness.

At the same time, there exists a dearth of sleep medicine specialists within the MHS, and demand for sleep specialty care greatly exceeds available supply.

Thus, the proposed study has direct military relevance because OSA telehealth care, if found effective, could be disseminated throughout the military as an evidence-based, cost-effective, broad-reaching, and convenient treatment approach to increase access to care. Hence this project is very timely, highly innovative, and scientifically sound, with great potential to enhance military telehealth efforts.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-64 years
2. ADFM or DEERS beneficiary
3. Enrolled in any TRICARE (Prime, Standard, or Extra)
4. Deferred to private sector care (i.e., local TRICARE network) for OSA care
5. Newly diagnosed with OSA (AHI>5)
6. Access to smartphone, desktop, laptop, or tablet computer

Exclusion Criteria:

1. History of prior OSA testing, diagnosis, or care
2. Contraindication for home sleep apnea testing, based on established AASM criteria
3. History of or high-risk for organic sleep disorders other than OSA (e.g., REM behavior disorder, obesity hypoventilation syndrome)
4. Active alcohol or substance dependence
5. Severe sleepiness (Epworth Sleepiness Scale [ESS]>18, or clinician judgment)
6. Pending permanent family change of station (PCS) within 6 months
7. Active-duty military service members (ADSM)
8. Untreated major medical or psychiatric illness
9. Pursuit of non-PAP treatment for OSA

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Apnea-Hypopnea Index (AHI): Assesses OSA severity via events/hour from diagnostic testing. | Participants are actively involved in the study for at least 90 days (approximately 3 months) following the initiation of PAP therapy.
  Unit: Events/hour
  Scale: Continuous; higher values = more severe outcome
Oxygen Desaturation Metrics: Reports oxygen nadir (%) and % of sleep time with saturation <90%. | Participants are actively involved in the study for at least 90 days (approximately 3 months) following the initiation of PAP therapy
  Units: Nadir (%), Time <90% (% of total sleep time)
  Scale: Continuous; lower nadir = worse outcome, higher time <90% = worse outcome
Positive Airway Pressure (PAP) Adherence | Participants are actively involved in the study for at least 90 days (approximately 3 months) following the initiation of PAP therapy.
  Includes treatment start date and usage (hours/night, % nights/week). Units: Start date; usage = hours/night, % nights/week
  Scale: Hours/night (min 0), % nights/week (0-100%); higher values = better outcome
PSQI: Pittsburgh Sleep Quality Index | Participants are actively involved in the study for at least 90 days (approximately 3 months) following the initiation of PAP therapy
  Assesses sleep quality (0-21); higher = poorer sleep.
  Scale: 0 - no difficulty and 21 indicating severe difficulties
ISI: Insomnia Severity Index | Participants are actively involved in the study for at least 90 days (approximately 3 months) following the initiation of PAP therapy
  Rates insomnia severity (0-28); higher = worse.
  Scale: 15-21 moderate insomnia, 22-28 severe insomnia.
ESS - Epworth Sleepiness Scale | Participants are actively involved in the study for at least 90 days (approximately 3 months) following the initiation of PAP therapy
  Assesses daytime sleepiness (0-24); higher = worse.
  Scale: 11-12 mild, 13-15 moderate, 16-24 excessive sleepiness.
FOSQ: Functional Outcomes of Sleep Questionnaire | Participants are actively involved in the study for at least 90 days (approximately 3 months) following the initiation of PAP therapy
  Evaluates OSA-related functional impact; higher scores = better functioning.
  Scale: 4 - no difficulty, 3 - yes, a little difficulty, 2 - yes, moderate difficulty, 1 - yes, extreme difficulty.
SF-12 - Short-form 12 | Participants are actively involved in the study for at least 90 days (approximately 3 months) following the initiation of PAP therapy.
  Evaluates general health-related quality of life.
  Scale: The scoring yields two summary measures: the Physical Component Summary (PCS) and the Mental Component Summary (MCS).
  Interpretation of Scores:
  Norm-based scoring system will be used to interpret PCS and MCS scores, with a mean of 50 and a standard deviation of 10 in the general population.
  Scores above 50 indicate a better-than-average health-while scores below 50 suggest below-average health.
PHQ-8 - Patient Health Questionnaire 8 | Participants are actively involved in the study for at least 90 days (approximately 3 months) following the initiation of PAP therapy.
  PHQ-8: Measures depressive symptoms (0-24); higher = worse.
  Scale: 0-4 no significant depression, 5-9 mild depressive symptoms, 10-14 moderate depressive symptoms, 15-19 moderately severe depressive symptoms, 20-24 severe depressive symptoms.
GAD-7: Generalized Anxiety Disorder - 7 | Participants are actively involved in the study for at least 90 days (approximately 3 months) following the initiation of PAP therapy
  Evaluates anxiety symptoms (0-21); higher = worse anxiety severity.
  Scale: 0-4 minimal anxiety, 5-9 mild anxiety, 10-14 moderate anxiety, 15-21 severe anxiety
PCL-5 - PTSD Checklist for DSM-5 | Participants are actively involved in the study for at least 90 days (approximately 3 months) following the initiation of PAP therapy.
  Evaluates trauma symptoms.
  Scale: 0-20 minimal symptoms, 21-40 mild symptoms, 41-60 moderate symptoms, 61-80 severe symptoms.
WPAI: Work Productivity and Activity Impairment Questionnaire | Participants are actively involved in the study for at least 90 days (approximately 3 months) following the initiation of PAP therapy
  Measures impairment in work/daily activities. Determines impact in percentages on absenteeism, presenteeism, overall work impairment, and activity impairment. higher %= greater impact.
  Scale: (0-100%), Higher scores indicate greater impairment and less productivity
RE-AIM: Reach, Effectiveness, Adoption, Implementation, Maintenance | Participants are actively involved in the study for at least 90 days (approximately 3 months) following the initiation of PAP therapy.
  Modified questionnaire to measure patient satisfaction. Formative evaluation
Health Care Utilization | Participants are actively involved in the study for at least 90 days (approximately 3 months) following the initiation of PAP therapy.
  Measures quantity healthcare services including dates and types of encounters, OSA diagnostic testing, and provision of PAP machines and supplies.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent F Capaldi II, M.D, Principal Investigator — Uniformed Services University Health Sciences
Locations (2):
- United States (2):
  - Uniformed Services University, Bethesda, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wickwire EM, Capaldi VF 2nd, So JY, Kim E, Thomas C, Johnston CW, Maggio S, Elmore JS, Albrecht JS, Verceles AC, Chen S. TELE-SLEEP OSA: A protocol for a hybrid type I randomized clinical trial of telemedicine for obstructive sleep apnea among military dependents and retirees. Contemp Clin Trials. 2026 Feb 4:108252. doi: 10.1016/j.cct.2026.108252. Online ahead of print. PMID 41651286